CLINICAL TRIAL: NCT05227794
Title: The Yale Equity in Student Well-Being Project: The Effects of 8-Week Online Compassion Cultivation Training (CCT) and Mindfulness-Based Stress Reduction (MBSR) on Diverse University Students' Social Well-Being and Mental Health
Brief Title: Compassion Training and Mindfulness Training for Social Well-Being and Mental Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2000031780
Record Dates: First submitted 2022-01-26; First posted 2022-02-07 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Anxiety; Depression; Stress; Burnout; Emotion Regulation; Social Acceptance; Loneliness; Compassion
Keywords: Mindfulness-Based Stress Reduction; Compassion Cultivation Training; Online Intervention; Undergraduate Students; Randomized Controlled Trial; Health Equity; Psychological Well-Being
MeSH Terms: conditions — Anxiety Disorders; Depression; Burnout, Psychological; Emotional Regulation; Psychological Well-Being | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: A three-arm randomized controlled trial will be conducted with eligible participants allocated to one of three parallel groups based on blinded randomization procedures (ratio of 1:1:1): 1) Compassion Cultivation Training (CCT), 2) Mindfulness-Based Stress Reduction (MBSR), and 3) Waitlist Control (WL). Randomization will take place after baseline assessment, so condition assignment does not influence pre-test data.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant Masking: Yes (partial)
  Participants will not be informed of the training they are randomly assigned. However, participants assigned to the waitlist will know they are in the control group (as they will not receive any training). Thus, comparisons between CCT and MBSR will be masked, but comparisons between CCT and MBSR with the control will not.
  Outcomes Assessor Masking: Yes (partial)
  For all self-reported outcomes (Primary Outcomes), partial participant blinding to condition will necessarily imply partial outcomes assessor blinding. Specifically, for CCT vs. MBSR comparisons, outcomes assessor blinding for self-reports will be masked, but comparisons between CCT and MBSR with the control will not be masked. For all peer rating outcomes (Other Outcomes), full outcomes assessor blinding will be possible (peers will not know what training group participants are in).
  Masking Conclusion:
  Double-blinding of the trial is possible (but see the above notes).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Compassion-Based Intervention (Experimental): Participants in this condition are assigned to an empirically supported 8-week online compassion-based intervention protocol. The intervention includes a weekly 2-hour educational session and a recommendation of 15-30-mins of daily meditation, and real-world assignments to practice compassion.
  Interventions: Behavioral: Compassion Cultivation Training (CCT)
- Mindfulness-Based Intervention (Experimental): Participants in this condition are assigned to an empirically supported 8-week online mindfulness-based intervention protocol. The intervention includes a weekly 2-hour educational session, a recommendation of 15-30 minutes of daily meditation, and an optional 6-hour one-day retreat.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction (MBSR)
- Waitlist Control (WL) (No Intervention): The WL control group will complete all study assessments on the same schedule as the intervention arms. At the time of the final follow-up assessment, participants will be randomly assigned to one of the interventions (CCT or MBSR) with the same instructors.

INTERVENTIONS:
Behavioral: Compassion Cultivation Training (CCT) — CCT is a secular, empirically supported 8-week program that integrates meditation practices, interactive discussions, and educational lectures to improve self-compassion and other-oriented compassion, emotion and stress management, and happiness and well-being. It includes a weekly 2-hour educational lecture with discussion and in-class exercises, a recommendation of 15-30 minutes of daily meditation, and real-world assignments to practice compassion. The program is taught by a certified instructor with more than 5 years experience.
  Other Names: CCT
  Arms: Compassion-Based Intervention
Behavioral: Mindfulness-Based Stress Reduction (MBSR) — MBSR is among the most studied mindfulness-based interventions in the literature and is a secular, 8-week psycho-educational group-based intervention. The program structure (slightly modified to match CCT) includes a weekly 2-hour class, a prescription of 15-30-minutes of daily mindfulness practice, and a one-day optional retreat (6 hours) between week six and seven. The program is taught by a certified instructor with more than 5 years experience.
  Other Names: MBSR
  Arms: Mindfulness-Based Intervention

SUMMARY:
Study Design, Aims, and Population:

The present study is a three-arm randomized controlled trial (RCT). The primary aim is to test the relative efficacy of two 8-week online interventions - Compassion Cultivation Training (CCT) and Mindfulness-Based Stress Reduction (MBSR) - in promoting diverse university students' social well-being (i.e., reduced loneliness, and enhanced social connectedness and perceived social support) compared to a Waitlist (WL) control group.

The secondary aim is to examine the effects of CCT versus MBSR on the mental health of diverse university students compared to the WL group. Mental health is defined in this research as both positive mental health (i.e., happiness, positive emotions, meaning and purpose) and negative mental health (i.e., stress, anxiety, and depression).

Additionally, another aim is to enroll 75% students of color and 50% male identifying students, whose social well-being and mental health is currently understudied, to better represent the sociodemographic diversity of the university student population in the literature.

Study Rationale:

The COVID-19 pandemic triggered widespread disruptions in social connections and relational bonds that robustly support a variety of mental and physical health-protective processes. University students' social well-being may have been especially impacted as universities provide a central context for socialization. At the same time, the pandemic exacerbated a pre-existing rise in cases of mental health conditions in university students. If found effective, online-based CCT and MBSR might serve as scalable psychological interventions to foster social thriving and mental health among diverse university students.

DETAILED DESCRIPTION:
Primary Aim and Hypotheses:

The primary aim is to study the main effects of CCT and MBSR (vs. WL, and compared to each other) on self-report measures of participant social well-being (i.e., loneliness, social connectedness, and perceived social support).

It is predicted that CCT will enhance social well-being compared to MBSR and to the WL, and that MBSR will enhance social well-being compared to the WL.

Secondary Aim and Hypotheses:

The secondary aim is to study the main effects of CCT and MBSR (vs. WL, and compared to each other) on self-report measures of participant mental health. This includes changes in positive mental health (i.e., happiness, positive emotions, and meaning and purpose) and negative mental health (i.e., stress, anxiety symptoms, and depression symptoms).

It is predicted that CCT and MBSR will both increase positive mental health and both decrease negative mental health compared to the WL. It is hypothesized that there will be no differences between the effects of CCT and MBSR on participants' positive or negative mental health.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled as a full-time Yale College undergraduate student

Exclusion Criteria:

* Current clinical mental health condition diagnosis made by a licensed medical professional (as self-reported by participants), including: major depressive disorder, anxiety disorder, bipolar disorder, borderline personality disorder, psychotic disorder, post-traumatic stress disorder, substance use disorder, and/or self-harm/attempted suicide/suicide ideation.

Demographic Eligibility Criteria:

* To enroll 75% participants of color (BIPOC) and 50% male identifying participants. Enrollment of participants who identify as White will be capped at n = 90, and participants who identify as female will be capped at n = 180.
* Participants will not be excluded based on any other demographic characteristics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Enrollment of participants who identify as female will be capped at n = 180 out N = 360 (50%).
Enrollment: 290 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Loneliness on the 4-point UCLA-Loneliness Scale Short-Form (LS-SF) at Week 10 (Post-Test) | Baseline and Week 10
  The UCLA LS-SF is a 10-item short-form to measure an individual's subjective feelings of loneliness and feelings of social isolation. Participants rate each item on a four-point scale ranging from 1 (I never feel this way) to 4 (I often feel this way).
  The UCLA LS-SF will be used as one measure out of three that will be aggregated into a single Social Well-Being Index (SWI) using latent variable modeling.
  Change = (Week 10 Score - Baseline Score)
Change from Baseline in Social Connectedness on the 6-point Social Connectedness Scale-Revised (SCS-R) at Week 10 (Post-Test) | Baseline and Week 10
  The 20-items SCS-R captures students' experience of closeness with others and maintaining and seeking connections. Sample items include "I am able to connect with other people," and "I am able to relate to my peers" "I see myself as a loner" and "I feel like an outsider." Items are rated on a six-point Likert-type scale ranging from 1 = "Strongly disagree" to 6 = "Strongly agree."
  The SCS-R will be used as one measure out of three that will be aggregated into a single Social Well-Being Index (SWI) using latent variable modeling.
  Change = (Week 10 Score - Baseline Score)
Change from Baseline in Perceived Social Support on the 5-point Medical Outcomes Study-Social Support Survey (MOS-SSS) at Week 10 (Post-Test) | Baseline and Week 10
  The MOS-SSS will be administered to measure perceived social support among college students (dropping the tangible support subscale due to lack of population relevance). Participants indicate their perceived level of current social support using a five-point Likert scale ranging from 1 (None of the time) to 5 (All of the time).
  The MOS-SSS will be used as one measure out of three that will be aggregated into a single Social Well-Being Index (SWI) using latent variable modeling.
  Change = (Week 10 Score - Baseline Score)

SECONDARY OUTCOMES:
Change from Baseline in Perceived Stress on the 5-point Perceived Stress Scale (PSS) at Week 10 (Post-Test) | Baseline and Week 10
  The 14-item PSS measures the degree to which situations in one's life are appraised as stressful. Respondents report how frequently they feel stress or have difficulty coping with life stresses. Items include questions that ask about the frequency of negative experiences (e.g., "In the last week, how often have you felt that you were unable to control the important things in your life?") and positive experiences (e.g., "In the last week, how often have you felt that things were going your way?"). Responses range from 0 = never to 4 = very often.
  The PSS will be used as one measure of three that will be aggregated into a single Negative Mental Health Index (NMHI) using latent variable modeling.
  Change = (Week 10 Score - Baseline Score)
Change from Baseline in Anxiety on the 5-point Patient-Reported Outcomes Measurement Information System Anxiety Short-Form (PROMIS-A-SF) at Week 10 (Post-Test) | Baseline and Week 10
  The PROMIS-A-SF is an 8-item measure to assess symptoms of anxiety among adults. The PROMIS anxiety items focus on fear and hyperarousal. The items in the PROMIS negative affect bank use a 7-day time frame and a five-point rating scale ranging from 1 (Never) to 5 (Always).
  The PROMIS-A-SF will be used as one measure of three that will be aggregated into a single Negative Mental Health Index (NMHI) using latent variable modeling.
  Change = (Week 10 Score - Baseline Score)
Change from Baseline in Depression on the 5-point Patient-Reported Outcomes Measurement Information System Depression Short-Form (PROMIS-D-SF) at Week 10 (Post-Test) | Baseline and Week 10
  The PROMIS-D-SF is an 8-item measure to assess symptoms of depression among adults. The PROMIS depression items focus on affective and cognitive manifestations of depression. The items in the PROMIS negative affect bank use a 7-day time frame and a five-point rating scale ranging from 1 (Never) to 5 (Always).
  The PROMIS-D-SF will be used as one measure of three that will be aggregated into a single Negative Mental Health Index (NMHI) using latent variable modeling.
  Change = (Week 10 Score - Baseline Score)
Change from Baseline in Happiness on the 7-point Subjective Happiness Scale (SHS) at Week 10 (Post-Test) | Baseline and Week 10
  The SHS is a 4-item scale that assesses global subjective happiness. One item asks respondents to characterize themselves on happiness using absolute ratings (1 = not a very happy person to 7 = a very happy person). Another item asks respondents to provide ratings of their happiness relative to their peers (1 = less happy to 7 = more happy). The final two items offer brief descriptions of happy and unhappy individuals and ask respondents the extent to which each characterization describes them (1 = not at all to 7 = a great deal). The 4 items are averaged with higher scores reflecting greater happiness (total score range: 1 = not at all happy to 7 = very happy).
  The SHS will be used as one measure of three that will be aggregated into a single Positive Mental Health Index (PMHI) using latent variable modeling.
  Change = (Week 10 Score - Baseline Score)
Change from Baseline in Positive Emotions on the 5-point Positive Emotions subscale of the Modified Differential Emotions Scale (mDES) at Week 10 (Post-Test) | Baseline and Week 10
  The Positive Emotions subscale of the Modified Differential Emotions Scale (mDES) measures the frequency one experiences 10 positive emotion word triads (e.g., 'serene-content-peaceful' and 'grateful-appreciative-thankful') 'over the past 2 weeks.' A composite score for positive emotions is created by averaging across the 10 positive emotion word triad items. Responses are made on a 5-point scale: 0 = never; 1 = rarely; 2 = some of the time; 3 = often; 4 = most of the time.
  The Positive Emotions subscale of the mDES will be used as one measure of three that will be aggregated into a single Positive Mental Health Index (PMHI) using latent variable modeling.
  Change = (Week 10 Score - Baseline Score)
Change from Baseline in Meaning and Purpose on the 5-point Patient-Reported Outcomes Measurement Information System Meaning and Purpose Scale Short-Form (PROMIS-MP-SF) at Week 10 (Post-Test) | Baseline and Week 10
  The Patient-Reported Outcomes Measurement Information System Meaning and Purpose Scale Short-Form (PROMIS-MP-SF) is comprised of four items. These four items are averaged to create a meaning and purpose mean score. The items are rated on a scale ranging from 1 (not at all) to 5 (very much).
  The PROMIS-MP-SF will be used as one measure of three that will be aggregated into a single Positive Mental Health Index (PMHI) using latent variable modeling.
  Change = (Week 10 Score - Baseline Score)

OTHER OUTCOMES:
Change from Baseline in Self-Compassion on the 5-point Self-Compassion-Scale (SCS) at Week 10 (Post-Test) | Baseline and Week 10
  The 26-item SCS assesses six aspects of Self-Compassion: Self-Kindness, Self-Judgment, Common Humanity, Isolation, Mindfulness, and Over-Identification. Responses are given on a five-point scale from 1 = "Almost Never" to 5 = "Almost Always."
  Change = (Week 10 Score - Baseline Score)
Change from Baseline in Other-Oriented Compassion on the 5-point Sussex Oxford Compassion Scale for Others (SOCS-O) at Week 10 (Post-Test) | Baseline and Week 10
  The SOCS-O is a validated 20-item self-report measure that assesses compassion for others based on five empirically supported elements: a) recognizing suffering; b) understanding the universality of suffering, c) feeling for the person suffering, d) tolerating uncomfortable feelings, and e) motivation to act/acting to alleviate suffering. Participants are asked how true each statement is, and responses are given on a five-point Likert scale, ranging from 1 (Not at all true) to 5 (Always true).
  Change = (Week 10 Score - Baseline Score)
Change from Baseline in Mindfulness on the 5-point Five-Facet Mindfulness Questionnaire-Short Form (FFMQ-SF) at Week 10 (Post-Test) | Baseline and Week 10
  The FFMQ-SF 24-item scale assesses five facets of a general tendency to be mindful in daily life: observing, describing, acting with awareness, nonreactivity to inner experience, and nonjudging of inner experience. Items are rated on a 5-point Likert-type scale ranging from 1 (never or very rarely true) to 5 (very often or always true).
  Change = (Week 10 Score - Baseline Score)
Change from Baseline in Emotion Regulation on the 5-point Cognitive Emotion Regulation Questionnaire (CERQ) at Week 10 (Post-Test) | Baseline and Week 10
  The Cognitive Emotion Regulation Questionnaire (CERQ) will be used to assess the strategies participants use to regulate their emotions. This measure includes 36 items that are rated on a scale from 1 (almost never) to 5 (almost always). This scale assesses multiple emotion regulation strategies, including 'maladaptive' emotion regulation strategies (e.g., rumination, catastrophizing) and 'adaptive' emotion regulation strategies (e.g., acceptance, positive reappraisal).
  Change = (Week 10 Score - Baseline Score)
Change from Baseline in Positive and Negative Affect on the 5-point Affective Experiences Scale (AES) at Week 10 (Post-Test) | Baseline and Week 10
  The Affective Experiences Scale (AES) assesses a wide range of positive and negative affective states using 48 single emotion word adjectives. The 48 items are aggregated into 16 three-item emotion word factors that assess affective experience (e.g., Pride = proud, accomplished, successful and Boredom = bored, disconnected, disengaged). Responses range from 1 = none of the time to 5 = all of the time.
  Change = (Week 10 Score - Baseline Score)
Change from Baseline in Discrimination-Based Trauma on the 4-point Trauma Symptoms of Discrimination Scale (TSDS) at Week 10 (Post-Test) | Baseline and Week 10
  The Trauma Symptoms of Discrimination Scale (TSDS) is a 21-item self-report scale that assesses anxiety-related trauma symptoms associated with experiences of discrimination. The TSDS is designed to assess lasting reactions to trauma from any kind of discrimination. Responses on the scale range from Never = 1 to Often = 4.
  Change = (Week 10 Score - Baseline Score)
Change from Baseline in Daily Social Well-Being on the Latent Factor-Scored Daily Social Well-Being Index (D-SWI) at Week 10 (Post-Test) | Baseline and Week 10
  A single Daily Social Well-Being Index (D-SWI) will be created with items from three scales (i.e., the UCLA Loneliness Scale-Short Form, the Social Connectedness Scale-Revised, and the Medical Outcomes Survey-Social Support Survey) using latent variable modeling. The D-SWI score will be a latent factor score produced by factor analysis.
  Using the daily diary method, assessments will occur daily from Baseline through Week 10.
  Change = Latent growth curve (LGC) of Baseline through Week 10 Scores
Change from Baseline in Daily Positive Mental Health on the Latent Factor-Scored Daily Positive Mental Health Index (D-PMHI) at Week 10 (Post-Test) | Baseline and Week 10
  A single Daily Positive Mental Health Index (D-PMHI) will be created with items from three scales (i.e., the Subjective Happiness Scale, the Modified Differential Emotions Scale-Positive Emotions Subscale, and the PROMIS Meaning and Purpose Scale) using latent variable modeling. The D-PMHI score will be a latent factor score produced by factor analysis.
  Using the daily diary method, assessments will occur daily from Baseline through Week 10.
  Change = Latent growth curve (LGC) of Baseline through Week 10 Scores
Change from Baseline in Daily Negative Mental Health on the Latent Factor-Scored Daily Negative Mental Health Index (D-NMHI) at Week 10 (Post-Test) | Baseline and Week 10
  A single Daily Negative Mental Health Index (D-NMHI) will be created with items from three scales (i.e., the Perceived Stress Scale, the PROMIS Anxiety Scale-Short Form, and the PROMIS Depression Scale-Short Form) using latent variable modeling. The D-NMHI score will be a latent factor score produced by factor analysis.
  Using the daily diary method, assessments will occur daily from Baseline through Week 10.
  Change = Latent growth curve (LGC) of Baseline through Week 10 Scores
Change from Baseline in Peer-Rated Social Well-Being on the Latent Factor-Scored Peer-Rated Social Well-Being Index (P-SWI) at Week 10 (Post-Test) | Baseline and Week 10
  A single Peer-Rated Social Well-Being Index (P-SWI) with items from three scales (i.e., the UCLA Loneliness Scale-Short Form, the Social Connectedness Scale-Revised, and the Medical Outcomes Survey-Social Support Survey) using latent variable modeling. The P-SWI score will be a latent factor score produced by factor analysis.
  Using the peer rating method, assessments will occur at Baseline and Week 10.
  Change = (Week 10 Factor Score - Baseline Factor Score)
Change from Baseline in Peer-Rated Positive Mental Health on the Latent Factor-Scored Peer-Rated Positive Mental Health Index (P-PMHI) at Week 10 (Post-Test) | Baseline and Week 10
  A single Peer-Rated Positive Mental Health Index (P-PMHI) will be created with items from three scales (i.e., the Subjective Happiness Scale, the Modified Differential Emotions Scale-Positive Emotions Subscale, and the PROMIS Meaning and Purpose Scale) using latent variable modeling. The P-PMHI score will be a latent factor score produced by factor analysis.
  Using the peer rating method, assessments will occur at Baseline and Week 10.
  Change = (Week 10 Factor Score - Baseline Factor Score)
Change from Baseline in Peer-Rated Negative Mental Health on the Latent Factor-Scored Peer-Rated Negative Mental Health Index (P-NMHI) at Week 10 (Post-Test) | Baseline and Week 10
  A single Peer-Rated Negative Mental Health Index (P-NMHI) will be created with items from three scales (i.e., the Perceived Stress Scale, the PROMIS Anxiety Scale-Short Form, and the PROMIS Depression Scale-Short Form) using latent variable modeling. The P-NMHI score will be a latent factor score produced by factor analysis.
  Using the peer rating method, assessments will occur at Baseline and Week 10.
  Change = (Week 10 Factor Score - Baseline Factor Score)
Change from Baseline in Social Well-Being on the Latent Factor-Scored Social Well-Being Index (SWI) at Week 22 (Post-Test) | Baseline and Week 22
  A single Social Well-Being Index (SWI) will be created from three scales (i.e., the UCLA Loneliness Scale-Short Form, the Social Connectedness Scale-Revised, and the Medical Outcomes Survey-Social Support Survey) using latent variable modeling. The SWI score will be a latent factor score produced by factor analysis.
  Assessments will occur at Baseline, Week 10, Week 14, and Week 22.
  Change = Latent growth curve (LGC) of Baseline, Week 10, Week 14, and Week 22 Scores
Change from Baseline in Positive Mental Health on the Latent Factor-Scored Positive Mental Index (PMHI) at Week 22 (Post-Test) | Baseline and Week 22
  A single Positive Mental Health Index (PMHI) will be created from three scales (i.e., the Subjective Happiness Scale, the Modified Differential Emotions Scale-Positive Emotions Subscale, and the PROMIS Meaning and Purpose Scale) using latent variable modeling. The PMHI score will be a latent factor score produced by factor analysis.
  Assessments will occur at Baseline, Week 10, Week 14, and Week 22.
  Change = Latent growth curve (LGC) of Baseline, Week 10, Week 14, and Week 22 Scores
Change from Baseline in Negative Mental Health on the Latent Factor-Scored Negative Mental Index (NMHI) at Week 22 (Post-Test) | Baseline and Week 22
  A single Negative Mental Health Index (NMHI) will be created from three scales (i.e., the Perceived Stress Scale, the PROMIS Anxiety Scale-Short Form, and the PROMIS Depression Scale-Short Form) using latent variable modeling. The NMHI score will be a latent factor score produced by factor analysis.
  Assessments will occur at Baseline, Week 10, Week 14, and Week 22.
  Change = Latent growth curve (LGC) of Baseline, Week 10, Week 14, and Week 22 Scores

CONTACTS AND LOCATIONS:
Overall Officials: Marc Brackett, PhD, Principal Investigator — Yale University; James Floman, PhD, Principal Investigator — Yale University
Locations (1):
- Yale Center for Emotional Intelligence, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lipson SK, Lattie EG, Eisenberg D. Increased Rates of Mental Health Service Utilization by U.S. College Students: 10-Year Population-Level Trends (2007-2017). Psychiatr Serv. 2019 Jan 1;70(1):60-63. doi: 10.1176/appi.ps.201800332. Epub 2018 Nov 5. PMID 30394183
- [Background] Wang X, Hegde S, Son C, Keller B, Smith A, Sasangohar F. Investigating Mental Health of US College Students During the COVID-19 Pandemic: Cross-Sectional Survey Study. J Med Internet Res. 2020 Sep 17;22(9):e22817. doi: 10.2196/22817. PMID 32897868
- [Background] Kirby JN. Compassion interventions: The programmes, the evidence, and implications for research and practice. Psychol Psychother. 2017 Sep;90(3):432-455. doi: 10.1111/papt.12104. Epub 2016 Sep 24. PMID 27664071
- [Background] Kirby JN, Tellegen CL, Steindl SR. A Meta-Analysis of Compassion-Based Interventions: Current State of Knowledge and Future Directions. Behav Ther. 2017 Nov;48(6):778-792. doi: 10.1016/j.beth.2017.06.003. Epub 2017 Jun 21. PMID 29029675
- [Background] Goldin, P. R., & Jazaieri, H. (2017). The compassion cultivation training (CCT) program. In E. M. Seppala, E. Simon-Thomas, S. L. Brown, M. C. Worline, C. D. Cameron, & J. R. Doty (Eds.), The Oxford Handbook of Compassion Science (pp. 235-245). Oxford University Press.
- [Background] Goldberg SB, Riordan KM, Sun S, Davidson RJ. The Empirical Status of Mindfulness-Based Interventions: A Systematic Review of 44 Meta-Analyses of Randomized Controlled Trials. Perspect Psychol Sci. 2022 Jan;17(1):108-130. doi: 10.1177/1745691620968771. Epub 2021 Feb 16. PMID 33593124
- [Background] Kabat-Zinn, J. (2003). Mindfulness-based stress reduction (MBSR). Constructivism in the Human Sciences, 8(2), 73.
- [Background] Kabat-Zinn, J. (2013). Full catastrophe living, revised edition: how to cope with stress, pain and illness using mindfulness meditation. Hachette, UK.
- [Background] Sedlmeier P, Eberth J, Schwarz M, Zimmermann D, Haarig F, Jaeger S, Kunze S. The psychological effects of meditation: a meta-analysis. Psychol Bull. 2012 Nov;138(6):1139-71. doi: 10.1037/a0028168. Epub 2012 May 14. PMID 22582738
- [Background] Sedlmeier, P., Loße, C. & Quasten, L.C. (2018). Psychological effects of meditation for healthy practitioners: an update. Mindfulness 9, 371-387. https://doi.org/10.1007/s12671-017-0780-4
- [Background] Sun S, Goldberg SB, Loucks EB, Brewer JA. Mindfulness-based interventions among people of color: A systematic review and meta-analysis. Psychother Res. 2022 Mar;32(3):277-290. doi: 10.1080/10503307.2021.1937369. Epub 2021 Jun 7. PMID 34098859
- [Background] Altman DG, Schulz KF, Moher D, Egger M, Davidoff F, Elbourne D, Gotzsche PC, Lang T; CONSORT GROUP (Consolidated Standards of Reporting Trials). The revised CONSORT statement for reporting randomized trials: explanation and elaboration. Ann Intern Med. 2001 Apr 17;134(8):663-94. doi: 10.7326/0003-4819-134-8-200104170-00012. PMID 11304107
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomized trials. Ann Intern Med. 2010 Jun 1;152(11):726-32. doi: 10.7326/0003-4819-152-11-201006010-00232. Epub 2010 Mar 24. PMID 20335313
- [Background] Bohlmeijer E, ten Klooster PM, Fledderus M, Veehof M, Baer R. Psychometric properties of the five facet mindfulness questionnaire in depressed adults and development of a short form. Assessment. 2011 Sep;18(3):308-20. doi: 10.1177/1073191111408231. Epub 2011 May 17. PMID 21586480
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Cella D, Riley W, Stone A, Rothrock N, Reeve B, Yount S, Amtmann D, Bode R, Buysse D, Choi S, Cook K, Devellis R, DeWalt D, Fries JF, Gershon R, Hahn EA, Lai JS, Pilkonis P, Revicki D, Rose M, Weinfurt K, Hays R; PROMIS Cooperative Group. The Patient-Reported Outcomes Measurement Information System (PROMIS) developed and tested its first wave of adult self-reported health outcome item banks: 2005-2008. J Clin Epidemiol. 2010 Nov;63(11):1179-94. doi: 10.1016/j.jclinepi.2010.04.011. Epub 2010 Aug 4. PMID 20685078
- [Background] Schalet BD, Pilkonis PA, Yu L, Dodds N, Johnston KL, Yount S, Riley W, Cella D. Clinical validity of PROMIS Depression, Anxiety, and Anger across diverse clinical samples. J Clin Epidemiol. 2016 May;73:119-27. doi: 10.1016/j.jclinepi.2015.08.036. Epub 2016 Feb 27. PMID 26931289
- [Background] Lyubomirsky, S., Lepper, H.S. A measure of subjective happiness: Preliminary reliability and construct validation. Social Indicators Research 46, 137-155 (1999). https://doi.org/10.1023/A:1006824100041
- [Background] Raes F, Pommier E, Neff KD, Van Gucht D. Construction and factorial validation of a short form of the Self-Compassion Scale. Clin Psychol Psychother. 2011 May-Jun;18(3):250-5. doi: 10.1002/cpp.702. Epub 2010 Jun 8. PMID 21584907
- [Background] Gu J, Baer R, Cavanagh K, Kuyken W, Strauss C. Development and Psychometric Properties of the Sussex-Oxford Compassion Scales (SOCS). Assessment. 2020 Jan;27(1):3-20. doi: 10.1177/1073191119860911. Epub 2019 Jul 29. PMID 31353931
- [Background] Lee, R. M., Draper, M., & Lee, S. (2001). Social connectedness, dysfunctional interpersonal behaviors, and psychological distress: Testing a mediator model. Journal of Counseling Psychology, 48(3), 310-318. https://doi.org/10.1037/0022-0167.48.3.310
- [Background] Mattick RP, Clarke JC. Development and validation of measures of social phobia scrutiny fear and social interaction anxiety. Behav Res Ther. 1998 Apr;36(4):455-70. doi: 10.1016/s0005-7967(97)10031-6. PMID 9670605
- [Background] Elphinstone, B. (2018). Identification of a Suitable Short-form of the UCLA-Loneliness Scale. Australian Psychologist, 53(2), 107-115. https://doi.org/10.1111/ap.12285
- [Background] Sherbourne CD, Stewart AL. The MOS social support survey. Soc Sci Med. 1991;32(6):705-14. doi: 10.1016/0277-9536(91)90150-b. PMID 2035047
- [Background] Jazaieri, H., Jinpa, G. T., McGonigal, K., Rosenberg, E. L., Finkelstein, J., Simon-Thomas, E., ... & Goldin, P. R. (2013). Enhancing compassion: A randomized controlled trial of a compassion cultivation training program. Journal of Happiness Studies, 14(4), 1113-1126. https://10.1007/s10902-012-9373-z
- [Background] Jazaieri, H., Lee, I. A., McGonigal, K., Jinpa, T., Doty, J. R., Gross, J. J., & Goldin, P. R. (2016). A wandering mind is a less caring mind: Daily experience sampling during compassion meditation training. The Journal of Positive Psychology, 11(1), 37-50. https://doi.org/10.1080/17439760.2015.1025418
- [Background] Fredrickson, B. L. (2013). Positive emotions broaden and build. Advances in Experimental Social Psychology, 47, 1-53. http://dx.doi.org/10.1016/ B978-0-12-407236-7.00001-2
- [Background] Williams, M. T., Printz, D., & DeLapp, R. C. T. (2018). Assessing racial trauma in African Americans with the Trauma Symptoms of Discrimination Scale. Psychology of Violence, 8, 735-747. doi:10.1037/vio0000212
- [Background] Garnefski, N., & Kraaij, V. (2006). Cognitive Emotion Regulation Questionnaire: Development of a short 18-item version (CERQ-Short). Personality and Individual Differences, 41, 1045-1053. doi:10.1016/j.paid.2006.04.010
- [Background] Salsman JM, Schalet BD, Park CL, George L, Steger MF, Hahn EA, Snyder MA, Cella D. Assessing meaning & purpose in life: development and validation of an item bank and short forms for the NIH PROMIS(R). Qual Life Res. 2020 Aug;29(8):2299-2310. doi: 10.1007/s11136-020-02489-3. Epub 2020 Apr 19. PMID 32306302
- [Background] Floman, J. L., Brackett, M., & Ponnock (2021) The Affective Experiences Scale (AES). Unpublished. Yale University.
- See also: Compassion Cultivation Training — https://www.compassioninstitute.com